CLINICAL TRIAL: NCT01285414
Title: A Phase 2 Study of Verubulin With Radiation Therapy and Temozolomide in Subjects Newly Diagnosed With Glioblastoma Multiforme
Brief Title: Verubulin, Radiation Therapy, and Temozolomide to Treat Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Myrexis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPC-6827-021
Record Dates: First submitted 2011-01-14; First posted 2011-01-28 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma; Brain Neoplasms; Brain Cancer; Verubulin
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — verubulin; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Verubulin & standard of care (RT & TMZ) (Experimental): Verubulin, at the dose selected in Part A, plus standard of care Radiation Therapy and Temozolomide
  Interventions: Drug: Verubulin
- Standard of care (RT & TMZ) (Active Comparator): Standard of care Radiation Therapy and Temozolomide
  Interventions: Drug: Temozolomide & Radiation Therapy

INTERVENTIONS:
Drug: Verubulin — Verubulin, dose determined in Part A, i.v. once weekly, Temozolomide & Radiation Therapy
  Other Names: Azixa; MPC-6827
  Arms: Verubulin & standard of care (RT & TMZ)
Drug: Temozolomide & Radiation Therapy — Temozolomide & Radiation Therapy
  Other Names: Temodar; TMZ; Radiotherapy
  Arms: Standard of care (RT & TMZ)

SUMMARY:
This, international, multi-center, Phase 2 study of verubulin will be conducted in patients with newly diagnosed Glioblastoma Multiforme (GBM). The study will be conducted in two parts. Part A is an open-label dose finding study that will determine the safety and tolerability of verubulin in combination with standard treatment. Part B is a randomized open-label study that will investigate progression-free survival and overall survival of patients receiving verubulin, at the dose determined in Part A, in combination with standard treatment versus standard treatment alone.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically proven, newly diagnosed glioblastoma multiforme
2. Age ≥ 18 years and < 70 years
3. Have an ECOG performance score of 0, 1, or 2, or KPS ≥ 70
4. Have adequate bone marrow function , liver function, and kidney function before starting therapy
5. Begin study therapy no more than 6 weeks after surgery or biopsy
6. Subjects that have had surgery must have an MRI ≤ 72 hours after surgery

Exclusion Criteria:

1. Have a carmustine implant (e.g., Gliadel® Wafer)
2. Have uncontrolled hypertension (SBP > 140 mmHg or DBP > 90 mmHg for more than 1 week)
3. Have a left ventricular ejection fraction below the lower limit of the reference range for the institution, as measured by multiple gated acquisition (MUGA) or echocardiogram (ECHO)
4. Have Troponin-I or Troponin T at Screening visit elevated above the upper limit of the reference range of the local institution
5. Have an increasing steroid requirement, indicative of a rapidly progressive disease
6. Have evidence of new, active intra tumor hemorrhage ≥ CTCAE Grade 2
7. Have had prior cranial radiotherapy
8. Have history of stroke and/or transient ischemic attack within 2 years of screening
9. Have history of cardiovascular disease (e.g., angina, myocardial infarction, congestive heart failure, etc.) within 2 years of screening
10. Be pregnant or breast feeding
11. Have a history of hypersensitivity reaction to Cremophor® EL
12. Have a history of hypersensitivity reaction or intolerance to temozolomide or dacarbazine (DTIC)

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Part A: Safety | 14 weeks
  Assess the number and percentage of subjects with adverse events, abnormal laboratory parameters, and ECG changes as measures of safety and tolerability.
Part B: 9 Mo Progression-free survival | 9 Month

SECONDARY OUTCOMES:
Part A: Pharmacokinetic Parameters | 18 weeks
  Measure the amount of verubulin in the body at specific time points when given with standard of care Radiation Therapy and Temozolomide
Part B: 6 Mo Progression Free Survival | 6 month
  Assess 6-month progression-free survival and compare median progression-free survival time for Radiation Therapy plus Temozolomide (TMZ)plus verubulin to standard of care (Radiation Therapy plus TMZ alone)
Overall Survival | 18 months
  Assess overall survival and compare median overall survival time for Radiation Therapy plus Temozolomide (TMZ)plus verubulin to standard of care (Radiation Therapy plus TMZ alone)
Part B: 12 Mo Progression Free Survival | 12 months
  Assess 12-month progression-free survival and compare median progression-free survival time for Radiation Therapy plus Temozolomide (TMZ)plus verubulin to standard of care (Radiation Therapy plus TMZ alone)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Beelen, MD, Study Director — Myrexis Inc.
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - University of Texas Health Science Center at Houston, Houston, Texas

REFERENCES:
- [Background] Sirisoma N, Pervin A, Zhang H, Jiang S, Willardsen JA, Anderson MB, Mather G, Pleiman CM, Kasibhatla S, Tseng B, Drewe J, Cai SX. Discovery of N-(4-methoxyphenyl)-N,2-dimethylquinazolin-4-amine, a potent apoptosis inducer and efficacious anticancer agent with high blood brain barrier penetration. J Med Chem. 2009 Apr 23;52(8):2341-51. doi: 10.1021/jm801315b. PMID 19296653
- [Background] Kasibhatla S, Baichwal V, Cai SX, Roth B, Skvortsova I, Skvortsov S, Lukas P, English NM, Sirisoma N, Drewe J, Pervin A, Tseng B, Carlson RO, Pleiman CM. MPC-6827: a small-molecule inhibitor of microtubule formation that is not a substrate for multidrug resistance pumps. Cancer Res. 2007 Jun 15;67(12):5865-71. doi: 10.1158/0008-5472.CAN-07-0127. PMID 17575155
- [Background] Tsimberidou AM, Akerley W, Schabel MC, Hong DS, Uehara C, Chhabra A, Warren T, Mather GG, Evans BA, Woodland DP, Swabb EA, Kurzrock R. Phase I clinical trial of MPC-6827 (Azixa), a microtubule destabilizing agent, in patients with advanced cancer. Mol Cancer Ther. 2010 Dec;9(12):3410-9. doi: 10.1158/1535-7163.MCT-10-0516. PMID 21159616
- See also: Additional Information — http://www.myrexis.com